CLINICAL TRIAL: NCT01191606
Title: Pressure-controlled Versus Volume-controlled Ventilation During Protective One Lung Ventilation for Thoracic Surgery
Brief Title: Pressure-controlled Versus Volume-controlled Ventilation During Protective One Lung Ventilation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Fellow, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: B-1005-100-003
Record Dates: First submitted 2010-08-05; First posted 2010-08-31 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-05

CONDITIONS: Arterial Oxygenation During Protective One Lung Ventilation
Keywords: pressure controlled; volume controlled; arterial oxygenation; one lung ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): the exchange of ventilatory mode from volume controlled ventilation to pressure controlled ventilation
  Interventions: Procedure: the change of ventilatory mode
- Group B (Active Comparator): the exchange of ventilatory mode from pressure controlled ventilation to volume controlled ventilation
  Interventions: Procedure: the change of ventilatory mode

INTERVENTIONS:
Procedure: the change of ventilatory mode — One lung ventilation initiated with volume controlled ventilation(OLV-VCV) with an inspired oxygen fraction (FIO2) of 1.0, a tidal volume 6 mL/kg based on PBW and respiratory rate to maintain PaCO2 between 35-45 mmHg. After 30 min, the ventilator was switched to pressure controlled ventilation and the inspiratory pressure was adjusted to obtain the tidal volume 6 mL/kg. No external positive end-expiratory pressure was applied throughout the entire study. Arterial PaO2, PaCO2, peak inspiratory pressure (Ppeak), mean inspiratory pressure (Pmean), plateau inspiratory pressure (Pplateau) were recorded at the end of each ventilaroty mode.
  Other Names: VCV-PCV group
  Arms: Group A
Procedure: the change of ventilatory mode — One lung ventilation initiated with pressure controlled ventilation with an inspired oxygen fraction (FIO2) of 1.0, an inspiratory pressure provided the tidal volume 6 mL/kg based on PBW and respiratory rate to maintain PaCO2 between 35-45 mmHg. After 30 min, the ventilator was switched to VCV with a tidal volume 6 mL/kg based on PBW. No external positive end-expiratory pressure was applied throughout the entire study. Arterial PaO2, PaCO2, peak inspiratory pressure (Ppeak), mean inspiratory pressure (Pmean), plateau inspiratory pressure (Pplateau) were recorded at the end of each ventilaroty mode.
  Other Names: PCV-VCV group
  Arms: Group B

SUMMARY:
The aim of this study is to determine the effects of pressure controlled ventilation during protective one lung ventilation on blood gases, airway pressures and hemodynamic variables compared with volume controlled ventilation.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) during thoracic surgery, in particular, video-assisted thoracic surgery is a standard practice to facilitate surgical exposure, but arterial hypoxemia has been a serious complication during one lung ventilation. Furthermore, recent studies have shown that one lung ventilation with a conventional tidal volume can involve lung injury associated with alveolar overdistension and high airway pressure. Therefore, lung protective ventilation with a low tidal volume during one lung ventilation has been suggested, and a recent study showed that protective ventilation during lung cancer surgery was associated with improved postoperative respiratory outcomes such as reduced incidence of acute lung injury and atelectasis.

During protective one lung ventilation limiting airway pressure and using low tidal volume, it is important to provide uniform alveolar expansion and maintain adequate oxygenation. A previous study suggested that the decelerating inspiratory flow delivery used in pressure controlled ventilation improved ventilation/perfusion distribution and arterial oxygenation during one lung ventilation5. Moreover, according to a recent study during laparoscopic obesity surgery, pressure-controlled ventilation improved oxygenation compared with volume controlled ventilation, which was associated with higher instantaneous flow peaks and a better alveolar recruitment6. On the other hand, other studies showed that ventilatory mode during one lung ventilation did not affect arterial oxygenation. However, these studies were performed during mechanical ventilation using conventional tidal volume, and the effect of ventilatory mode during protective one lung ventilation on oxygenation has not been clearly determined yet.The aim of this study is to determine the effects of pressure controlled ventilation during protective one lung ventilation on blood gases, airway pressures and hemodynamic variables compared with volume controlled ventilation.

ELIGIBILITY:
Inclusion Criteria:

* patients (ASA physical status I-III) undergoing elective thoracic surgery in the lateral position with at least 1 h of one lung ventilation

Exclusion Criteria:

* patients with major organ dysfunction, hemodynamic instability, or increased intracranial pressure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
arterial oxygenation differences | four time points during operation
  (1) during two-lung ventilation using VCV before initiation of OLV (baseline); (2) during OLV 30 min after the first randomized ventilation mode; (3) 30 min after the second ventilation mode; and (4) 30 min after reestablishing two-lung ventilation.

SECONDARY OUTCOMES:
peak inspiratory pressure (Ppeak) | four time points during operation
  (1) during two-lung ventilation using VCV before initiation of OLV (baseline); (2) during OLV 30 min after the first randomized ventilation mode; (3) 30 min after the second ventilation mode; and (4) 30 min after reestablishing two-lung ventilation.
mean inspiratory pressure (Pmean) | four time points during operation
  (1) during two-lung ventilation using VCV before initiation of OLV (baseline); (2) during OLV 30 min after the first randomized ventilation mode; (3) 30 min after the second ventilation mode; and (4) 30 min after reestablishing two-lung ventilation.
plateau inspiratory pressure (Pplateau) | four time points during operation
  (1) during two-lung ventilation using VCV before initiation of OLV (baseline); (2) during OLV 30 min after the first randomized ventilation mode; (3) 30 min after the second ventilation mode; and (4) 30 min after reestablishing two-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Young Hwang, MD, Principal Investigator — Fellow
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea